CLINICAL TRIAL: NCT05335889
Title: Feasibility of Using Wearable Sensors and Artificial Intelligence for Carbohydrate Counting in Chinese Americans With Type 2 Diabetes
Brief Title: Wearable Sensors and Artificial Intelligence for Carbohydrate Counting
Status: Completed | Type: Observational
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Other Study IDs: 21-01714
Record Dates: First submitted 2022-03-10; First posted 2022-04-20 (Actual); Last update posted 2024-04-12 (Actual); Status verified 2024-04

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Continuous Glucose Monitoring

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Type 2 Diabetes group: Participants with Type 2 Diabetes will wear eButton and Continuous Glucose Monitoring (CGM) for 2 weeks and complete food diaries to record carb grams.
  Interventions: Device: eButton; Device: Continuous Glucose Monitoring (CGM)

INTERVENTIONS:
Device: eButton — The eButton is a wearable camera that takes pictures every 6 seconds of whatever is in front of participants. The recorded data are processed by algorithms to determine food names, volumes, and nutrient value of the consumed food (e.g., grams of carbohydrates). The eButton is a wearable device containing a multicore microprocessor, a rechargeable battery capable of 10-15 hours of continuous operation (upon a flexible choice of battery capacity), a miniSD card for data storage.
Device: Continuous Glucose Monitoring (CGM) — The use of this device provides ambulatory glucose profiles, giving graphic and quantitative information on 24-hour glucose patterns. It does not require finger-prick testing for calibration. The system consists of a reader and a sensor (35 mm x 5 mm). The sensor is applied to the back of a person's arm. The sensor automatically measures interstitial glucose at 15-minute intervals during daily activities like work, sleep, eating, and exercise. It is able to store blocks of glucose data for 14 days.
  Other Names: FreeStyle Libre Pro model

SUMMARY:
This is a one-group pilot study where Chinese immigrants who are English speaking with T2D from NYU Langone Health and NYU Brooklyn Family Health Center (Sunset Park) will be recruited.

DETAILED DESCRIPTION:
To evaluate the estimation accuracy using eButton, researchers will collect carbohydrate data via weighing food by registered dietitian nutritionist (RDN) ("gold standard") (2 days/week at research labs) and food diaries by participants (2 days/week at research labs and 3 days/ week at participant home). Then, the estimated carb grams will be compared head to head among each other. Assessment will be at 0 and 2 weeks, including surveys and qualitative audio interview.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years old
* Diagnosed with T2D at least one year prior
* Self-identified as first- or second-generation Chinese immigrants
* Feel comfortable communicating in English, the reason is that the questionnaires/surveys are validated in English
* Have a computer and internet connection

Exclusion Criteria:

* Plan frequent travel or vacations or plan to relocate in the next five weeks
* Have serious diabetes-related complications, physical illness, or mental illness (e.g., schizophrenia, bipolar disorder, or substance abuse) that would preclude participation
* Have severe cognitive impairments (e.g., dementia, intellectual disability)

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Chinese Americans participants are targeted to test eButton accuracy is that most Chinese Americans live closely within the community (e.g., Chinatown) and use a handful of Asian stores as their main food sources, which reduces the complexity of their food choices. Thus, collecting data from this ethnic group can provide an in-depth validation of eButton closed-loop feedback concept without excessive experimental time.
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2022-07-18 (Actual); Primary Completion 2023-09-22 (Actual); Study Completion 2023-09-22 (Actual)

PRIMARY OUTCOMES:
Accuracy of Carbohydrate Counting using eButton (absolute error) | Day 14
  The estimated carb grams using the eButton, gold standard, and participants' food diaries will be compared head to head among each other. The absolute error will be computed: the difference between the estimated value and the gold standard (estimated - gold standard). Bland-Altman plots will be used to examine the level of agreement between eButton and gold standard measurements.
Accuracy of Carbohydrate Counting using eButton (relative error) | Day 14
  The estimated carb grams using the eButton, gold standard, and participants' food diaries will be compared head to head among each other. The relative error will be computed: the percentage difference between the estimated value relative to the gold standard. Relative errors will be reported using boxplots to allow visual comparison of the distribution and variability in errors across all methods. Bland-Altman plots will be used to examine the level of agreement between eButton and gold standard measurements.
Proportion of participants who are fully compliant with eButton use | Day 14
  Proportion of participants who are fully compliant with eButton use and proportion of meals evaluated using eButton, with 95% confidence intervals will be qualitatively reported. Perceived usefulness and perceived ease of use will be summarized as mean and standard deviation.

CONTACTS AND LOCATIONS:
Overall Officials: Yaguang Zheng, PhD, RN, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research
Access Criteria: The investigator who proposed to use the data. Upon reasonable request. Requests should be directed to yaguang.zheng@nyu.edu. To gain access, data requestors will need to sign a data access agreement.

DOCUMENTS (1):
  • Informed Consent Form (2022-05-23): https://cdn.clinicaltrials.gov/large-docs/89/NCT05335889/ICF_000.pdf